CLINICAL TRIAL: NCT00208104
Title: Motivational Interviewing in Hypertensive African Americans
Brief Title: Motivational Interviewing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AAAA0311; R01HL069408-03 (NIH); NCT00201175 (obsolete NCT alias)
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Essential Hypertension
Keywords: Hypertension; African Americans; Adherence; Motivational Interviewing
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interview Condition (Experimental): Trained nurses will interview the group using motivational interview counseling techniques. All sessions will be conducted with the aid of an adapted version of a standardized structured adherence counseling script. This script was specifically developed for use in medication adherence studies of HIV positive patients and has been provided for this trial.
  Interventions: Behavioral: Motivational Interviewing
- Non-supportive Counseling (No Intervention): A non-supportive counseling session will consist of regular nurse-patient interaction.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Trained nurses will interview the group using motivational interview counseling techniques. All sessions will be conducted with the aid of an adapted version of a standardized structured adherence counseling script. This script was specifically developed for use in medication adherence studies of HIV positive patients and has been provided for this trial.
  Arms: Motivational Interview Condition

SUMMARY:
The purpose of this project is to study ways to make it more likely that patients will take their blood pressure medicine as recommended by their doctors.

DETAILED DESCRIPTION:
The objective of this randomized control trial is to evaluate, among 190 African-American patients with poorly controlled hypertension followed in a community-based primary care practice, whether motivational interviewing is more effective than usual care (routine counseling) in achieving adherence to prescribed blood pressure medications at 12 months.

The project aims to: 1) determine whether patients who receive motivational interview counseling have greater reduction in both systolic and diastolic blood pressure than those in the control group at 12 months. Clinic blood pressure readings will be assessed at baseline and at every three months thereafter for one year and 2) assess the effect of self-efficacy and intrinsic motivation as potential mediators of motivational interview on adherence. Self-efficacy and intrinsic motivation will be assessed at baseline and every three months thereafter for one year.

ELIGIBILITY:
Inclusion Criteria:

The target population consisted of hypertensive African American patients who fulfilled the following eligibility criteria:

* Self-identification as African American
* Age 18 years or older
* Diagnosis of hypertension utilizing ICD-9 codes 401-401.9 (the code for essential hypertension)
* Taking at least one antihypertensive medication
* Uncontrolled hypertension of a clinic blood pressure reading >140/90 mm Hg or 130/80 mm Hg (for those with kidney disease or diabetes) on two successive clinic visits prior to screening (defined per JNC VI criteria)
* Fluent in English language

Exclusion Criteria:

Participants were excluded if they:

* Had a diagnosis of cognitive impairment or serious medical condition as determined by their primary physician
* Were unable to give informed consent
* Refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2002-07; Primary Completion 2006-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Score on Morisky Medication Adherence Scale (MMAS-4) | Up to one year from baseline
  Adherence to antihypertensive medications will be assessed at baseline and every three months thereafter for one year using a validated 4-item scale developed by Morisky that specifically addresses medication-taking. The scale asks patients to respond "yes" or "no" to a set of 4 questions. A positive response to any question indicates a problem with adherence. Each positive answer is assigned a score of 1. The total possible score is 4 with higher score indicating poorer adherence.

SECONDARY OUTCOMES:
Blood pressure readings | Up to one year from baseline
  Within clinic systolic and diastolic blood pressure readings will be assessed at baseline and at every three months thereafter for one year using a mercury syphgmomanometer.
Score on efficacy scale | Up to one year from baseline
  Self-efficacy will be assessed at baseline and every three months thereafter for one year using a 44-item self-efficacy scale devised based on Bandura's Scale. Patients are asked to rate their confidence in taking their blood pressure medications under a variety of situations that may pose difficulties to them using a 3-point likert response format - 1= not at all sure, 2= somewhat sure, and 3= very sure. A summary score is computed by summing the responses, with higher scores reflecting high self-efficacy.
Score on the Treatment Self-Regulation Questionnaire (TSRQ) | Up to one year from baseline
  Intrinsic motivation will be assessed at baseline and every three months thereafter for one year with aid of TSRQ. It is used to assess the degree to which one's motivation for a particular behavior is relatively autonomous or self-determined. Patients are provided with 15 reasons why they may not take their medications as prescribed and asked to indicate the degree to which each reason is true on a scale of 1 to 7 with 7 been very true.

CONTACTS AND LOCATIONS:
Overall Officials: Gbenga Ogedegbe, MD, MS, MPH, Principal Investigator — CUMC
Locations (1):
- Columbia University Medical Center, New York, New York, United States